CLINICAL TRIAL: NCT02745236
Title: The Effect of Nurse Practitioner-Led Care on Health Related Quality Of Life in Adult Patients With Atrial Fibrillation - A Randomized Trial
Brief Title: The Effect of Nurse Practitioner Led-Care on Quality of Life in Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University Hospital Foundation (Other)
Responsible Party: Principal Investigator, Marcie Smigorowsky, PhD Student Faculty of Medicine and Dentistry, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: MSmig01
Record Dates: First submitted 2016-04-16; First posted 2016-04-20 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Health Related Quality of Life; Nurse Practitioner; Sustainable Models of Healthcare; Patient Satisfaction
MeSH Terms: conditions — Atrial Fibrillation; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse Practitioner Led-Care (Experimental): Nurse Practitioner (NP) Intervention Initial Visit and Interventions: An experienced nurse practitioner with extra atrial fibrillation (AF) management training will complete the initial assessment to determine a treatment plan based on current AF Guidelines. The NP will provide patient education on AF management.
  Follow-up: Follow-up will occur at 3 and 6 months from baseline to evaluate the patient's response to treatment and will be modified as required based on AF symptoms, testing results and physical assessment.
  A physician will be consulted for advanced specialty AF management or if a patient requires admission to hospital.
  Interventions: Other: Nurse Practitioner Led-Care
- Cardiologist Led-Care (Active Comparator): Standard Care Initial Visit and Intervention: A general cardiologist will manage patients as per their usual practice.
  Follow-up: As per the cardiologist's usual practice. The patient's care will remain with the family physician if no follow-up is required.
  Follow-up: Follow-up will be determined as per the cardiologist's usual practice. If a follow-up appointment is required it will done in the cardiologist's own independent clinic. The patient's care will be referred back to the family physician if no follow-up is required.
  Interventions: Other: Cardiologist Led-Care

INTERVENTIONS:
Other: Nurse Practitioner Led-Care — Diagnosis and treatment plan decisions will be determined by Nurse Practitioner Led-Care.
  Other Names: Intervention Arm
  Arms: Nurse Practitioner Led-Care
Other: Cardiologist Led-Care — Diagnosis and treatment plan decisions will be determined as per usual care by the Cardiologist
  Other Names: Control Arm
  Arms: Cardiologist Led-Care

SUMMARY:
Atrial fibrillation (AF) is the most common heart rhythm disease characterized by an irregular heart rhythm of the top part (atria) of the heart. It may cause unpleasant symptoms as well as increases the person's risk of stroke and heart failure. With an ageing population, increasing rates of AF and limited access to specialists, new methods of care, like nurse practitioners (NP) need to be assessed to meet patient specific needs and provide sustainable care.

The objective of the project is to evaluate the effect of Nurse Practitioner-led care in people with AF on their quality of life.

The Canadian Healthcare system is overwhelmed, with increasing costs and wait times. Contributing to these issues, is AF is the most common arrhythmia accompanied with costly complications including stroke and heart failure. Currently family or emergency room physicians ask general cardiologists or specialized cardiologists, to provide care to patients with AF. Unfortunately, there is limited access to their services. NP's are nurses who have taken extra education at University to treat patients and prescribe medications. This research project involves an NP who has specialized training in AF patient management.

By utilizing an NP to provide care for patients with AF, the investigators hope to improve patient's quality of life and satisfaction with care. This may also reduce complications of AF.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Documented non valvular atrial fibrillation
* Able to provide informed consent
* Able and willing to complete the study questionnaires on own or with assistance

Exclusion Criteria:

* Referral is for atrioventricular node ablation or pulmonary vein isolation.
* Patients who have failed antiarrhythmic medications
* Patients with moderate to severe mitral or aortic valvular heart disease
* Clinically unstable atrial fibrillation
* Cannot or unwilling to attend follow-up appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-07-31 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Difference in change in Atrial Fibrillation Effect on Quality of Life (AFEQT) scores between groups | At 6 months

SECONDARY OUTCOMES:
Difference in change in EQ-5D scores between groups | At 6 months
Difference in composite outcomes of death from cardiovascular causes, cardiovascular hospitalization and emergency room visits between groups | At 6 months
Satisfaction with NP-led or cardiologist care as measured by the overall mean score of the Consultant Satisfaction Questionnaire (CSG). | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcie J Smigorowsky, PhD, NP, Principal Investigator — University of Alberta; Ross T Tsuyuki, PharmD, MSc, Principal Investigator — University of Alberta
Locations (1):
- Mazankowski Alberta Heart Institution, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cairns JA, Healey JS, Macle L, Mitchell LB, Verma A; Canadian Cardiovascular Society Atrial Fibrillation Guidelines Committee. The new Canadian Cardiovascular Society algorithm for antithrombotic therapy of atrial fibrillation is appropriately based on current epidemiologic data. Can J Cardiol. 2015 Jan;31(1):20-3. doi: 10.1016/j.cjca.2014.11.021. Epub 2014 Nov 26. No abstract available. PMID 25547545
- [Background] Verma A, Cairns JA, Mitchell LB, Macle L, Stiell IG, Gladstone D, McMurtry MS, Connolly S, Cox JL, Dorian P, Ivers N, Leblanc K, Nattel S, Healey JS; CCS Atrial Fibrillation Guidelines Committee. 2014 focused update of the Canadian Cardiovascular Society Guidelines for the management of atrial fibrillation. Can J Cardiol. 2014 Oct;30(10):1114-30. doi: 10.1016/j.cjca.2014.08.001. Epub 2014 Aug 13. PMID 25262857
- [Background] Faxon DP, Schwamm LH, Pasternak RC, Peterson ED, McNeil BJ, Bufalino V, Yancy CW, Brass LM, Baker DW, Bonow RO, Smaha LA, Jones DW, Smith SC Jr, Ellrodt G, Allen J, Schwartz SJ, Fonarow G, Duncan P, Horton K, Smith R, Stranne S, Shine K; American Heart Association's Expert Panel on Disease Management. Improving quality of care through disease management: principles and recommendations from the American Heart Association's Expert Panel on Disease Management. Circulation. 2004 Jun 1;109(21):2651-4. doi: 10.1161/01.CIR.0000128373.90851.7B. No abstract available. PMID 15173048
- [Background] Campbell DJ, Sargious P, Lewanczuk R, McBrien K, Tonelli M, Hemmelgarn B, Manns B. Use of chronic disease management programs for diabetes: in Alberta's primary care networks. Can Fam Physician. 2013 Feb;59(2):e86-92. PMID 23418263
- [Background] Gillis AM, Burland L, Arnburg B, Kmet C, Pollak PT, Kavanagh K, Veenhuyzen G, Wyse DG. Treating the right patient at the right time: an innovative approach to the management of atrial fibrillation. Can J Cardiol. 2008 Mar;24(3):195-8. doi: 10.1016/s0828-282x(08)70583-x. PMID 18340388
- [Background] Ross H, Higginson LA, Ferguson A, O'Neill BJ, Kells CM, Cox JL, Sholdice MM. Too many patients, too few cardiologists to care? Can J Cardiol. 2006 Sep;22(11):901-2. doi: 10.1016/s0828-282x(06)70308-7. No abstract available. PMID 17016884
- [Background] Kinnersley P, Anderson E, Parry K, Clement J, Archard L, Turton P, Stainthorpe A, Fraser A, Butler CC, Rogers C. Randomised controlled trial of nurse practitioner versus general practitioner care for patients requesting "same day" consultations in primary care. BMJ. 2000 Apr 15;320(7241):1043-8. doi: 10.1136/bmj.320.7241.1043. PMID 10764366
- [Background] Seale C, Anderson E, Kinnersley P. Comparison of GP and nurse practitioner consultations: an observational study. Br J Gen Pract. 2005 Dec;55(521):938-43. PMID 16378563
- [Background] Thrasher C, Purc-Stephenson R. Patient satisfaction with nurse practitioner care in emergency departments in Canada. J Am Acad Nurse Pract. 2008 May;20(5):231-7. doi: 10.1111/j.1745-7599.2008.00312.x. PMID 18460162
- [Background] Oliver GM, Pennington L, Revelle S, Rantz M. Impact of nurse practitioners on health outcomes of Medicare and Medicaid patients. Nurs Outlook. 2014 Nov-Dec;62(6):440-7. doi: 10.1016/j.outlook.2014.07.004. Epub 2014 Aug 1. PMID 25172368
- [Background] Hendriks JM, de Wit R, Crijns HJ, Vrijhoef HJ, Prins MH, Pisters R, Pison LA, Blaauw Y, Tieleman RG. Nurse-led care vs. usual care for patients with atrial fibrillation: results of a randomized trial of integrated chronic care vs. routine clinical care in ambulatory patients with atrial fibrillation. Eur Heart J. 2012 Nov;33(21):2692-9. doi: 10.1093/eurheartj/ehs071. Epub 2012 Mar 27. PMID 22453654
- [Background] Johnston BC, Patrick DL, Busse JW, Schunemann HJ, Agarwal A, Guyatt GH. Patient-reported outcomes in meta-analyses--Part 1: assessing risk of bias and combining outcomes. Health Qual Life Outcomes. 2013 Jul 1;11:109. doi: 10.1186/1477-7525-11-109. PMID 23815754
- [Background] Spertus J, Dorian P, Bubien R, Lewis S, Godejohn D, Reynolds MR, Lakkireddy DR, Wimmer AP, Bhandari A, Burk C. Development and validation of the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire in patients with atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):15-25. doi: 10.1161/CIRCEP.110.958033. Epub 2010 Dec 15. PMID 21160035
- [Background] Dorian P, Cvitkovic SS, Kerr CR, Crystal E, Gillis AM, Guerra PG, Mitchell LB, Roy D, Skanes AC, Wyse DG. A novel, simple scale for assessing the symptom severity of atrial fibrillation at the bedside: the CCS-SAF scale. Can J Cardiol. 2006 Apr;22(5):383-6. doi: 10.1016/s0828-282x(06)70922-9. PMID 16639472
- [Background] Dorian P, Guerra PG, Kerr CR, O'Donnell SS, Crystal E, Gillis AM, Mitchell LB, Roy D, Skanes AC, Rose MS, Wyse DG. Validation of a new simple scale to measure symptoms in atrial fibrillation: the Canadian Cardiovascular Society Severity in Atrial Fibrillation scale. Circ Arrhythm Electrophysiol. 2009 Jun;2(3):218-24. doi: 10.1161/CIRCEP.108.812347. Epub 2009 Mar 31. PMID 19808471
- [Background] Baker R. Development of a questionnaire to assess patients' satisfaction with consultations in general practice. Br J Gen Pract. 1990 Dec;40(341):487-90. PMID 2282225
- [Background] Poulton BC. Use of the consultation satisfaction questionnaire to examine patients' satisfaction with general practitioners and community nurses: reliability, replicability and discriminant validity. Br J Gen Pract. 1996 Jan;46(402):26-31. PMID 8745848
- [Background] Bungard TJ, Smigorowsky MJ, Lalonde LD, Hogan T, Doliszny KM, Gebreyesus G, Garg S, Archer SL. Cardiac EASE (Ensuring Access and Speedy Evaluation) - the impact of a single-point-of-entry multidisciplinary outpatient cardiology consultation program on wait times in Canada. Can J Cardiol. 2009 Dec;25(12):697-702. doi: 10.1016/s0828-282x(09)70530-6. PMID 19960130
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Derived] Smigorowsky MJ, Norris CM, McMurtry MS, Tsuyuki RT. Measuring the effect of nurse practitioner (NP)-led care on health-related quality of life in adult patients with atrial fibrillation: study protocol for a randomized controlled trial. Trials. 2017 Aug 3;18(1):364. doi: 10.1186/s13063-017-2111-4. PMID 28774317